CLINICAL TRIAL: NCT04152811
Title: Cooking Matters for Diabetes - Practical Application of Diabetes Self-Management Education
Brief Title: Cooking Matters for Diabetes - A 6-Week Program for Practical Application of Diabetes Self-Management Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Principal Investigator, Joshua Joseph, MD, Assistant Professor of Medicine, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019H0095
Record Dates: First submitted 2019-08-21; First posted 2019-11-05 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus; Type 1 Diabetes; Type 2 Diabetes
Keywords: nutrition; cooking; diabetes self-management education
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Waitlist Control Design
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Waitlist 1 (Active Comparator): usual diabetes care
  Interventions: Other: Usual Diabetes Care
- Intervention 1 (Experimental): 6-weeks of cooking matters for diabetes classes
  Interventions: Behavioral: Cooking Matters for Diabetes
- Waitlist 2 (Active Comparator): usual diabetes care
  Interventions: Other: Usual Diabetes Care
- Intervention 2 (Experimental): 6-weeks of cooking matters for diabetes classes
  Interventions: Behavioral: Cooking Matters for Diabetes

INTERVENTIONS:
Behavioral: Cooking Matters for Diabetes — Each Cooking Matters course is made up of 6, 2-hour, weekly classes with 15 participants. The curricula is based on the Dietary Guidelines for Americans, MyPlate, the American Diabetes Association Standards of Medical Care in Diabetes 2017 and Medical Nutrition Therapy Evidence Based Guide for Practice/Nutrition Protocol as the foundation for basic nutrition guidelines, then builds upon these ideas using the collective groups' needs and interest to provide interactive lessons to teach cooking, food safety and food resource management with emphasis placed on blood sugar management.
  Arms: Intervention 1; Intervention 2
Other: Usual Diabetes Care — Usual Diabetes Care
  Arms: Waitlist 1; Waitlist 2

SUMMARY:
Our primary objective is to improve glycemic control (Hemoglobin A1c [HbA1c]) over 3 months in individuals with diabetes by teaching practical application of diabetes education through "Cooking Matters" compared to usual care.

Our secondary objective is to improve health related quality of life, adherence to diabetes self-management behaviors (physical activity, diet, glucose monitoring, and medication adherence) over 3-months compared to usual care.

We hypothesize that participants in the cooking matters intervention will have significant improvement in glycemic control (HbA1c), HRQOL, and adherence to diabetes self- management compared to usual care. Our study is significant as it examines a novel approach to improving diabetes care and addressing glycemic control in diabetes.

DETAILED DESCRIPTION:
We will enroll 60 participants with diabetes and HbA1c ≥ 7% in a Cooking Matters (CM) program using a waitlist control design with 30 participants in the intervention group and 30 participants in the waitlist control group, separated into two arms.Participants will be stratified by sex and randomized using a random number generator program to either the intervention or wait list control group. Each CM course is made up of 6, 2-hour, weekly classes with 15 participants. The curricula is based on the Dietary Guidelines for Americans, MyPlate (the current nutrition guide published by the USDA Center for Nutrition Policy and Promotion, a food circle depicting a place setting with a plate and glass divided into five food groups), the American Diabetes Association Standards of Medical Care in Diabetes 2017 and Medical Nutrition Therapy Evidence Based Guide for Practice/Nutrition Protocol as the foundation for basic nutrition guidelines, then builds upon these ideas using the collective groups' needs and interest to provide interactive lessons to teach cooking, food safety and food resource management with emphasis placed on blood sugar management. Five of the 6 classes will include hands-on cooking instruction and nutrition instruction; one of the 6 classes will be a grocery store tour held in a grocery store of the groups' choosing. This class will provide nutrition instruction with the focus on meal planning for optimal glucose control under the constraints of a budget. Each class will be interactive and provides participants opportunities to demonstrate their understanding of the lesson. Participants are encouraged to ask questions, offer solutions and share their experiences. At the end of each class, when food preparation is highlighted, the class and instructors will gather to sample all recipes and have open discussion. Each participant will take home a bag of groceries with the ingredients to replicate the recipes made in class. At the beginning of each class, participants are encouraged to share with the group how they used of the previous week's groceries and reflect on cooking at home. We will administer validated surveys measuring health-related quality of life, diabetes self-management behaviors, and dietary patterns and perform point of care HbA1c assessment of both groups (intervention and waitlist control) when intervention 1 begins the program in week 1. We will then proceed with the CM intervention with intervention 1 in weeks 1 thru 6 and the post test will be administered to the intervention group at the end of the intervention, 3, 6 and 12 months post intervention. In week 18-23, we will administer CM to the original waitlist control group and they will follow the same protocol as intervention 1. The second arm of the study will follow the same design, beginning in week 12 of the study.

ELIGIBILITY:
Inclusion criteria

* Interest in cooking education for diabetes
* Diagnosis of diabetes
* Prior diabetes education
* Most recent HbA1c ≥ 7%
* Appropriate for a group class setting

Exclusion Criteria

* Previous participation in Cooking Matters program
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c over 4.5 months | Change in Hemoglobin A1c from baseline (0 months) to 4.5 months
  Change in Hemoglobin A1c over 4.5 months

SECONDARY OUTCOMES:
Change in Health Related Quality of Life over 4.5 months using SF-12 Survey | Change in Health Related Quality of Life from baseline (0 months) to 4.5 months using SF-12 Survey
  Change in Health Related Quality of Life over 4.5 months using SF-12 Survey

CONTACTS AND LOCATIONS:
Overall Officials: Joshua J Joseph, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center - Outpatient Care East, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams A, Shrodes JC, Radabaugh JN, Braun A, Kline D, Zhao S, Brock G, Nolan TS, Garner JA, Spees CK, Joseph JJ. Outcomes of Cooking Matters for Diabetes: A 6-week Randomized, Controlled Cooking and Diabetes Self-Management Education Intervention. J Acad Nutr Diet. 2023 Mar;123(3):477-491. doi: 10.1016/j.jand.2022.07.021. Epub 2022 Aug 10. PMID 35961614
- [Derived] Shrodes JC, Williams A, Nolan TS, Radabaugh JN, Braun A, Kline D, Zhao S, Brock G, Garner JA, Spees CK, Joseph JJ. Feasibility of Cooking Matters for Diabetes: A 6-week Randomized, Controlled Cooking and Diabetes Self-Management Education Intervention. J Acad Nutr Diet. 2023 Mar;123(3):492-503.e5. doi: 10.1016/j.jand.2022.07.020. Epub 2022 Aug 6. PMID 35944873